CLINICAL TRIAL: NCT03158467
Title: A Pilot Randomized Control Trial of Advance Care Planning and Triggered Palliative Care for Cancer Patients Undergoing Stem Cell Transplantation (RCT of ACP for Transplant)
Brief Title: RCT of ACP for Transplant
Status: Withdrawn | Type: Observational
Why Stopped: Did not enroll
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: UPCC 23417
Record Dates: First submitted 2017-05-16; First posted 2017-05-18 (Actual); Last update posted 2018-09-20 (Actual); Status verified 2018-05

CONDITIONS: Cancer Patients Undergoing Stem Cell Transplantation (RCT of ACP for Transplant)
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Phase 1
  Interventions: Other: Surveys
- Phase 2
  Interventions: Other: Surveys

INTERVENTIONS:
Other: Surveys — Instruments will be administered via the online RedCAP platform. The survey instruments will include a Decision Conflict Scale (DCS), the McGill Quality of Life (MQoL), the Human Connection (THC), and a general demographics questionnaire. Patients will have the opportunity to complete the instruments via a research iPad while in clinic or via a survey link emailed to their private email account.

SUMMARY:
We aim to examine the effect of an online advance directive on decisional conflict and quality of life in patients undergoing stem cell transplant. We also aim to assess the effect of palliative care at the time of a sentinel event on quality of life.

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria for Phase I (primary objective) are as follows:

* Age ≥ 18 years
* Hematologic malignancy diagnosis including any subset of myeloma, lymphoma, leukemia, or myelodysplastic syndrome
* Currently scheduled for autologous or allogeneic transplant at the Hospital of the University of Pennsylvania

The inclusion criteria for Phase II (secondary objective) are as follows:

* Age ≥ 18 years
* Hematologic malignancy diagnosis including any subset of lymphoma, leukemia, or myelodysplastic syndrome
* Received an autologous or allogeneic stem cell transplant at the Hospital of the University of Pennsylvania and experienced a sentinel event of either 1) disease relapse,2) severe (Grade III or IV) graft-versus-host disease, or 3) unplanned hospital admission with length of stay greater than 72 hours.

Exclusion Criteria:

The exclusion criteria for Phase I include:

* Inability to read and write English
* Not serving as the primary decision maker for their health-related decisions
* Having a non-hematologic malignancy reason for undergoing transplantation (e.g. aplastic anemia)

The exclusion criteria for Phase II include:

* Not completing participation in Phase I of the study
* Myeloma diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer Patients Undergoing Stem Cell Transplantation
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2019-05-15 (Estimated); Study Completion 2019-11-15 (Estimated)

PRIMARY OUTCOMES:
Number of surveys completed | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Pallavi Kumar, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine